CLINICAL TRIAL: NCT01750996
Title: Strongest Families Finland Canada: Family-based Prevention and Treatment Program of Early Childhood Disruptive Behavior
Acronym: Fin-Can
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIHR# 103146
Record Dates: First submitted 2011-11-14; First posted 2012-12-17 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Disruptive Behavior Disorder
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care control (Parenting tips) (No Intervention): Participants randomized to usual care will have access to a brief information website containing brief parenting tips but will not receive Strongest Families Intervention
- Strongest Families (Experimental): Strongest Families intervention
  Interventions: Behavioral: Strongest Families

INTERVENTIONS:
Behavioral: Strongest Families — Behavioural intervention
  Arms: Strongest Families

SUMMARY:
The goal of the Strongest Families Finland Canada project is to help parents develop skills to strengthen their families and reduce disruptive behavior in their 4 year old children.

DETAILED DESCRIPTION:
This project will have two phases, described below. The first part will be development of the web based program, the second part will be the implementation of the program in Finland. All participants will be recruited in Finland and all research activities will take place in Finland, by the Finnish Consortium. The Canadian Consortium will assist in funding and provide expert support.

Part 1: Website development:

The Strongest families program provides evidence based psychological and behavioural interventions to families with children with mild to moderate mental health problems. Parents work through a handbook with exercises, watch instructional videos and participate in weekly phone calls from a trained 'coach' (paraprofessional) to provide support, respond to parents' questions and highlight the skills included in a handbook. The preliminary analysis of a Strongest Families effectiveness trial based at the Izaak Walton Killam Children's Hospital (IWK) Health Centre (Projects #2234, and #2654) and effect size reports from the IWK Strongest families Service Program suggest that Strongest Families is an effective treatment for Oppositional Defiant Disorder (ODD).

Strongest Families is an adaptation of the COPE program. COPE is a large-group parent training program (average 25 families per group) that has been evaluated and used in many centres across Canada, the United States and Europe. It was developed at McMaster University by a team led by Dr. Charles Cunningham (one of the investigators on this submission). The groups use a coping modelling problem solving approach to skill acquisition which encourages parents to discuss the solution to common problems, collaborate in the formulation of child management strategies, share successes, and provide supportive feedback. Large group discussions may also provide more information regarding normal child development and a greater perspective on common child management difficulties than clinic/individual parent training .

The benefits for parents participating in COPE group sessions are many, but the burden of traveling to receive services can impede attendance, especially for families in rural areas. One solution to this issue would be to adapt individualized Strongest Families to a more accessible mode.

We propose to develop a web-based version of Strongest Families in preparation for a Randomized Control Trial (RCT) in Finland. All components of web site will be developed using a collaborative approach with active participation by all members of the research team. We will review each of the component as it is developed. We estimate a minimum of three rounds of testing for each component. The program will be evaluated using the user-interface so that we review the website and all its various features in a manner that simulates the actual parent experience. No qualitative or quantitative data will be recorded for this phase of the project. No participants will be recruited for this phase of the trial.

The web version of Strongest Families will have two components. First, is a personalized website that tracks and uses all activities and interactions to modify the Strongest Families intervention as the user progresses through the sessions. Interactions include questions, surveys, and polls which will be asked periodically throughout the program (for examples see Appendix A). Second, the parenting skills curriculum will be based on our Strongest Families program, an approach derived from programs developed by members of this team18,19. Third, parents , using pseudonyms, will participate in a discussion board/blog to exchange ideas. Pseudonyms will be chosen by the participant, but will not include any identifying elements.

Part 2: Randomized trial (Conducted in Finland, no Canadian recruitment)

The centerpiece project will be a population-based RCT of high risk 4 year olds attending well-child clinics in Turku and environs. Families of children with behavioural challenges fort he last six months, scoring 5 points or more on the Conduct subscale of the Strengths and Difficulties Questionnaire (SDQ) and with some perceived problems by the parent in the impact section of the SDQ will be offered participation in a 2 arm trial. All data will be collected in Finland and stored at the University of Turku. All forms/scripts/ measures will be administered in Finnish or Swedish. This project has been approved by the Intermunicipal Hospital District of Southwest Finland. The Canadian team will provide expert and financial support.

Treatment Group: Families randomized to Web-Enhanced Strongest Families (described above) will receive the website program described above.

Control Group: Families randomized to Educational Control will receive access to a static website with parenting tips as well as a 45 coaching call to review the parenting tips.

Randomization: (1:1 treatment: control; stratified by sex). Randomization sequences were generated by a qualified expert at arms length to the trial using a random permuted block sequence generator then concealed the placements using a double envelop system labeled with sequential numbers. Study staff were blinded to placements until randomization was completed by a study staff delegate.

ELIGIBILITY:
Inclusion Criteria:

* Child is 4 years old at time of recruitment
* Parent/guardian has access to a computer and the internet
* Parent/guardian is comfortable reading at a Grade 5 level
* Child meets screening criteria (SDQ score of 4 or more with some problems per impact score)

  * Child has had behavioural challenges for the last 6 months
  * Parent has access to phone in home
  * Parent speaks/writes Finnish

Exclusion Criteria:

* - Has received or is receiving behavioral treatment (parent training) before
* Diagnosis of:

  * Autism or a Pervasive development disorder (PDD)
  * Down's syndrome
  * Fetal Alcohol Syndrome
  * Mental retardation
  * Genetic diagnosis that will lead to mental retardation
  * Major mental health disorder (e.g., depression, psychosis)
* Child is not speaking using a sentence
* Child is deaf or blind

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
CHild Behaviour Checklist (to measure change from baseline) | Measure change from baseline at 6 & 12 months
  Measure of child behavioural change from baseline to 6 & 12 months

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale Short Form (DASS-21)- Finnish | Baseline, 6 & 12months
  Parental stress changes from baseline will be measured over time
The Parenting Scale (To measure change from baseline to 6 & 21 months) | To measure change from baseline to 6 & 12 months post randomization
  Measure parental parenting practice changes from baseline
Barkley's Quick-Screen: The Barkley Adult ADHD Rating Scale IV (to measure change from baseline) | Measure change from baseline to 6&12 months
  To measure parental ADHD symptom changes form baseline
Child Behaviour Checklist- Teacher version (to measure change since baseline) | Measure change from Baseline to 6 & 12 months
  To measure child behaviour changes at daycare from baseline to 6 & 12 months post randomization
Satisfaction measure: Researcher designed for the Intervention group | end of program intervention (average is about 5 months but timing of completion varies between participants.)
  To measure satisfaction with Intervention and website information
Strengths & Difficulties Questionnaire (Screening Tool) | Screening
  Screening tool used to identify high risk 4 year olds
The Parent Problem Checklist | Measure change from Baseline to 6 & 12 months
  To measure interparental conflict
The Sense of Coherence Scale (SOC-13) | Measure change from Baseline to 6 & 12 months
  To measure parent's sense of coherence (i.e., global view of the world, and individual environment as comprehensible, manageable and meaningful)
The Inventory of Callous-Unemotional Traits | Measure change from Baseline to 6 & 12 months
  To measure child empathy

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- University of Turku, Finland, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Aggregate summary data would be made available but not individual data.

REFERENCES:
- [Background] McGrath PJ, Sourander A, Lingley-Pottie P, Ristkari T, Cunningham C, Huttunen J, Filbert K, Aromaa M, Corkum P, Hinkka-Yli-Salomaki S, Kinnunen M, Lampi K, Penttinen A, Sinokki A, Unruh A, Vuorio J, Watters C. Remote population-based intervention for disruptive behavior at age four: study protocol for a randomized trial of Internet-assisted parent training (Strongest Families Finland-Canada). BMC Public Health. 2013 Oct 21;13:985. doi: 10.1186/1471-2458-13-985. PMID 24139323
- [Result] Sourander A, McGrath PJ, Ristkari T, Cunningham C, Huttunen J, Lingley-Pottie P, Hinkka-Yli-Salomaki S, Kinnunen M, Vuorio J, Sinokki A, Fossum S, Unruh A. Internet-Assisted Parent Training Intervention for Disruptive Behavior in 4-Year-Old Children: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Apr;73(4):378-87. doi: 10.1001/jamapsychiatry.2015.3411. PMID 26913614
- [Derived] Rissanen E, Kuvaja-Kollner V, Kankaanpaa E. Cost-Effectiveness of Digital Preventive Parent Training for Early Childhood Disruptive Behaviour. J Ment Health Policy Econ. 2024 Sep 1;27(3):85-98. PMID 39290059
- [Derived] Sourander A, Ristkari T, Kurki M, Gilbert S, Hinkka-Yli-Salomaki S, Kinnunen M, Pulkki-Raback L, McGrath PJ. Effectiveness of an Internet-Based and Telephone-Assisted Training for Parents of 4-Year-Old Children With Disruptive Behavior: Implementation Research. J Med Internet Res. 2022 Apr 4;24(4):e27900. doi: 10.2196/27900. PMID 35377332
- [Derived] Sourander A, McGrath PJ, Ristkari T, Cunningham C, Huttunen J, Hinkka-Yli-Salomaki S, Kurki M, Lingley-Pottie P. Two-Year Follow-Up of Internet and Telephone Assisted Parent Training for Disruptive Behavior at Age 4. J Am Acad Child Adolesc Psychiatry. 2018 Sep;57(9):658-668.e1. doi: 10.1016/j.jaac.2018.07.001. Epub 2018 Aug 3. PMID 30196869